CLINICAL TRIAL: NCT02349399
Title: Drug Utilization Study on Diane®-35 (and Generics) in European Healthcare Databases
Brief Title: Drug Utilization Study on Diane-35 (and Generics) in Three European Healthcare Databases
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 17660; DI1402 (Other: Company internal)
Record Dates: First submitted 2015-01-23; First posted 2015-01-28 (Estimated); Last update posted 2017-04-05 (Actual); Status verified 2017-04

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Cyproterone; Ethinyl Estradiol; Cyproterone acetate, ethinyl estradiol drug combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Drug Utilisation / Cohort 1: New users of CPA/EE in 2011/2012 and in 2014
  Interventions: Drug: Cyproterone / Ethinylestradiol (Diane-35, BAY86-5264) and its Generics

INTERVENTIONS:
Drug: Cyproterone / Ethinylestradiol (Diane-35, BAY86-5264) and its Generics — Hormonal Contraceptive: Cyproterone Acetate 2 mg / Ethinylestradiol 35 μg

SUMMARY:
The study objectives are to characterize new users of Cyproterone Acetate / Ethinylestradiol (CPA/EE) in 2011/2012 and in 2014 according to demographics, treatment characteristics, previous diagnosis of acne, hirsutism or other hyperandrogenic conditions, previous acne treatment and (concomitant) use of hormonal contraceptives identified in Healthcare Databases in the UK (THIN), the Netherlands (PHARMO) and Italy (HSD).

ELIGIBILITY:
Inclusion Criteria:

* The study population will include all female patients registered in the investigated healthcare databases receiving CPA/EE in 2011 or 2012 (first run) or 2014 (second run), without a prescription of CPA/EE in the year prior to index date. Only patients with recorded history in the database of ≥ 365 days prior to index date will be included in the study.

Exclusion Criteria:

* <365 days recorded history in the database prior to index date
* a prescription of CPA/EE in the year prior to index date

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women who are new users of CPA/EE in 2011/2012 and in 2014
Sampling Method: Non-Probability Sample
Enrollment: 26065 (Actual)
Dates: Start 2015-05-01 (Actual); Primary Completion 2016-03-01 (Actual); Study Completion 2016-03-01 (Actual)

PRIMARY OUTCOMES:
Proportion (%) of new users of Diane-35 (or generics) with a previous diagnosis of Acne | up to 12 months
Proportion (%) of new users of Diane-35 (or generics) with a previous diagnosis of Hirsutism | up to 12 months
Proportion (%) of new users of Diane-35 (or generics) with a previous diagnosis of other Hyperandrogenic Conditions (e.g. androgenic alopecia, seborrhea, polycystic ovary syndrome) | up to 12 months

SECONDARY OUTCOMES:
Determination of previous acne treatments (prescription drugs only) of Diane-35 (or generics) users with a previous diagnosis of acne. | up to 12 months
Proportion (%) of new Diane-35 (or generics) users, who have concomitant prescriptions of other combined oral contraceptives | up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (3):
- Many Locations, Italy
- Many Locations, Netherlands
- Many Locations, United Kingdom